CLINICAL TRIAL: NCT04056325
Title: Efficacy, Safety and Pharmacokinetics of Ascending Dosages of Moxidectin Alone and in Comparison to Ivermectin Against Strongyloides Stercoralis in Adults: a Randomized Controlled Trial
Brief Title: Efficacy, Safety, and PK of Ascending Dosages of Moxidectin Versus Ivermectin Against Strongyloides Stercoralis
Acronym: StrongMoxi
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: National Institute of Public Health, Vientiane, Laos (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Jennifer Keiser, PhD, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2019-07-22; First posted 2019-08-14 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Strongyloides Stercoralis Infection
MeSH Terms: interventions — moxidectin; Ivermectin

STUDY DESIGN:
Intervention Model Description: Phase 2a: Parallel study with 7 treatment arms (including a placebo arm) Phase 2b: Parallel study with 2 treatment arms
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Phase 2a: single-blinded (participant and lab technician) Phase 2b: double-blinded (participant, Care Provider) PK sub-studies are single-blinded (participant)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Phase 2a - Arm A (Experimental): 2 mg Moxidectin at day 0 administered orally
  Interventions: Drug: Moxidectin
- Phase 2a - Arm B (Experimental): 4 mg Moxidectin at day 0 administered orally
  Interventions: Drug: Moxidectin
- Phase 2a - Arm C (Experimental): 6 mg Moxidectin at day 0 administered orally
  Interventions: Drug: Moxidectin
- Phase 2a - Arm D (Experimental): 8 mg Moxidectin at day 0 administered orally
  Interventions: Drug: Moxidectin
- Phase 2a - Arm E (Experimental): 10 mg Moxidectin at day 0 administered orally
  Interventions: Drug: Moxidectin
- Phase 2a - Arm F (Experimental): 12 mg Moxidectin at day 0 administered orally
  Interventions: Drug: Moxidectin
- Phase 2a - Arm G (Placebo Comparator): matching Placebo tablet(s) at day 0 administered orally
  Interventions: Drug: Placebo oral tablet
- Phase 2b - Arm A (Experimental): the recommended dose moxidectin (i.e. the most promising dosage identified in phase 2a; between 2-12 mg) at day 0 administered orally
  + Ivermectin placebo, corresponding to Phase 2b - Arm B
  Interventions: Drug: Moxidectin
- Phase 2b - Arm B (Active Comparator): 200 µg/kg ivermectin at day 0 administered orally
  + Moxidectin placebo, corresponding to Phase 2b - Arm A
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Moxidectin — Monotherapy, oral administration, single dose, fixed dose
  Arms: Phase 2a - Arm A; Phase 2a - Arm B; Phase 2a - Arm C; Phase 2a - Arm D; Phase 2a - Arm E; Phase 2a - Arm F; Phase 2b - Arm A
Drug: Ivermectin — Monotherapy, oral administration, single dose, weight dependent
  Arms: Phase 2b - Arm B
Drug: Placebo oral tablet — Monotherapy, oral administration, single dose, matching number of tablets
  Arms: Phase 2a - Arm G

SUMMARY:
This study is a phase 2, blinded and randomized clinical trial. The phase 2a trial is single blinded and conducted in Lao, while the phase 2b trial is double-blinded and conducted in Lao and Cambodia. The study aims at providing evidence on effective doses and safety of moxidectin in adults against infection with S. stercoralis in Laos (trial 2a) and efficacy and safety of moxidectin compared to ivermectin in adults against infection with S. stercoralis in Laos and Cambodia (trial 2b). The efficacy of the treatment will be assessed by collecting three stool samples once pre-treatment and once 21 days post-treatment. The stool samples will be analyzed by a quantitative Baermann assay.

DETAILED DESCRIPTION:
This is a phase 2a single-blinded and a phase 2b double-blinded randomized clinical trial, which aims to determine efficacy and safety of (2a) seven ascending oral moxidectin dosages in 210 adults infected with S. stercoralis, namely placebo, 2 mg, 4 mg, 6 mg, 8 mg, 10 mg, 12 mg in Lao and (2b) the recommended dose moxidectin (i.e. the most promising dosage identified in trial A; between 2-12 mg) in comparison to the standard treatment dose of ivermectin (200 µg/kg) in 350 adults infected with S. stercoralis in Lao and Cambodia. Embedded in the trial is a pharmacokinetic/-dynamic study with the goal to measure moxidectin disposition in adults and to determine population pharmacokinetic (PK) parameters of the optimal dose of moxidectin in the treatment of S. stercoralis.

The primary objective is to determine the dose-response of moxidectin based on cure rates (CR) against S. stercoralis and to quantify the efficacy of the recommended dose to the standard treatment (ivermectin) in adults.

The secondary objectives of the trial are: Evaluation of the safety and tolerability of the dose-dependent treatment regimes, evaluation of the safety and tolerability of moxidectin compared to ivermectin, comparison of the larvae reduction rate (LRR) of the different treatment regimens against S. stercoralis (trial 2a,b), determination of an exposure- (including Cmax, area under curve (AUC) and tmax) -response correlation of moxidectin in adults, comparison of the exposure-response of moxidectin using venous and capillary blood, evaluation of the cure rate of the different moxidectin treatment regimens against co-infection and the determination of the population PK parameters of the optimal dose of moxidectin in the treatment of S. stercoralis.

After obtaining informed consent from each individual, the medical history of the participants will be assessed with a standardized questionnaire, in addition to a clinical examination carried out by the study physician before treatment. Enrollment will be based on collection and analysis by a quantitative Baermann method (in duplicates) of three stool samples. Randomization of participants into the different treatment arms will be stratified according to intensity of infection. The adults will also be interviewed before treatment, 3 and 24 hours as well as 21 days after treatment about the occurrence of adverse events (AE). The efficacy of the treatment will be determined 21 days post-treatment by collecting another three stool samples. All stool samples will be examined with duplicate Baermann assays recorded quantitatively. Co-infection with T. trichiura, A. lumbricoides and hookworm infection will be identified using duplicate Kato-Katz thick smears on stool samples.

A subsample of adults will further be sampled using finger pricking for micro sampling at 0, 2, 4, 8, 24, and 72 hours, 7 and 21 days post treatment to evaluate pharmacokinetic parameters (trial phase 2a) and at defined time windows, that are based on the PK model earned from trial 2a (trial phase 2b). For validation of the analytical method the subsample of one study arm (8 mg, trial phase 2a) will undergo venous blood sampling in addition to finger pricking.

An available case analysis (full analysis set according to the intention to treat principle) will be performed, including all subjects with primary end point data. Supplementary, a per-protocol analysis will be conducted. CRs will be calculated as the percentage of larvae-positive subjects at baseline who become larvae-negative after treatment. Larvae per gram (LPG) stool sample will be assessed by calculating the mean of the larvae counts from the three duplicate Baermann assays and divided by the mean weighted amount of these stool samples. The LRR will be calculated following: (LRR = (1-(mean at follow-up/mean at baseline))*100) Geometric and arithmetic mean larvae counts will be calculated for the different treatment arms before and after treatment to assess the corresponding LRRs. Bootstrap resampling method with 2,000 replicates will be used to calculate 95% confidence intervals (CIs) for LRRs. Emax models using the dose finding package of the statistical software environment R will be implemented to predict the dose-response curves in terms of CRs and LRRs.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years) infected with S. stercoralis
* Absence of major systemic illnesses
* Written informed consent signed by individual

Exclusion Criteria:

* Any abnormal medical conditions or chronic disease
* Negative diagnostic result for S. stercoralis
* No written informed consent by individual.
* Pregnant and lactating women.
* Recent use of anthelmintic drug (within past 4 weeks), attending other clinical trials during the study
* Known allergy to study medications (i.e. moxidectin, ivermectin)
* Currently taking medications with known interaction (i.e. for warfarin)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 617 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keiser, Prof. Dr., Principal Investigator — Swiss TPH
Locations (1):
- National Institute of Public Health, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sprecher VP, Hofmann D, Savathdy V, Xayavong P, Norkhankhame C, Huy R, Khieu V, Sayasone S, Hattendorf J, Keiser J. Efficacy and safety of moxidectin compared with ivermectin against Strongyloides stercoralis infection in adults in Laos and Cambodia: a randomised, double-blind, non-inferiority, phase 2b/3 trial. Lancet Infect Dis. 2024 Feb;24(2):196-205. doi: 10.1016/S1473-3099(23)00507-8. Epub 2023 Nov 7. PMID 37949090
- [Derived] Smit C, Hofmann D, Sayasone S, Keiser J, Pfister M. Characterization of the Population Pharmacokinetics of Moxidectin in Adults Infected with Strongyloides Stercoralis: Support for a Fixed-Dose Treatment Regimen. Clin Pharmacokinet. 2022 Jan;61(1):123-132. doi: 10.1007/s40262-021-01048-4. Epub 2021 Jul 23. PMID 34296417
- [Derived] Hofmann D, Sayasone S, Sengngam K, Chongvilay B, Hattendorf J, Keiser J. Efficacy and safety of ascending doses of moxidectin against Strongyloides stercoralis infections in adults: a randomised, parallel-group, single-blinded, placebo-controlled, dose-ranging, phase 2a trial. Lancet Infect Dis. 2021 Aug;21(8):1151-1160. doi: 10.1016/S1473-3099(20)30691-5. Epub 2021 Mar 30. PMID 33798487

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2a - Arm A (Moxidectin 2 mg): 2 mg Moxidectin at day 0 administered orally
- Phase 2a - Arm B (Moxidectin 4 mg): 4 mg Moxidectin at day 0 administered orally
- Phase 2a - Arm C (Moxidectin 6 mg): 6 mg Moxidectin at day 0 administered orally
- Phase 2a - Arm D (Moxidectin 8 mg): 8 mg Moxidectin at day 0 administered orally
- Phase 2a - Arm E (Moxidectin 10 mg): 10 mg Moxidectin at day 0 administered orally
- Phase 2a - Arm F (Moxidectin 12 mg): 12 mg Moxidectin at day 0 administered orally
- Phase 2a - Arm G (Placebo): matching Placebo tablet(s) at day 0 administered orally
- Phase 2b - Arm A (Moxidectin): 8 mg moxidectin (i.e. the most promising dosage identified in trial A; between 2-12 mg) at day 0 administered orally
  + Ivermectin placebo dose, corresponding to Phase 2b - Arm B
- Phase 2b - Arm B (Ivermectin): 200 µg/kg ivermectin at day 0 administered orally
  + Moxidectin placebo dose, corresponding to Phase 2b - Arm A
Period: Phase 2a
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Started | 31 | 33 | 33 | 32 | 32 | 30 | 32 | 0 | 0
Completed | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 0 | 0
Not Completed | 1 | 4 | 1 | 3 | 2 | 0 | 3 | 0 | 0
Period: Phase 2b
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 197 | 197
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 192 | 189
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Phase 2b - Arm A (Moxidectin): 8 mg moxidectin (i.e. the most promising dosage identified in phase 2a; between 2-12 mg) at day 0 administered orally
  + Ivermectin placebo dose, corresponding to Phase 2b - Arm B
- Total: Total of all reporting groups
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin) | Total
Number analyzed (Participants) | 31 | 33 | 33 | 32 | 32 | 30 | 32 | 197 | 197 | 617
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: In phase 2a, the analysis population is the intention-to-treat population, excluding participants lost to follow-up. In phase 2b, the analysis population includes all randomized participants.
  years
    number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 197 | 197 | 603
    (all) | 41.6 (10.7) | 46.3 (12.5) | 45.3 (11.8) | 44.0 (13.5) | 44.4 (11.8) | 44.3 (11.2) | 40.0 (10.7) | 45.4 (11.6) | 44.8 (11.1) | 45.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: In phase 2a, the analysis population is the intention-to-treat population, excluding participants lost to follow-up. In phase 2b, the analysis population includes all randomized participants.
  Participants
    number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 197 | 197 | 603
    Female | 12 | 8 | 10 | 9 | 13 | 9 | 10 | 89 | 94 | 254
    Male | 18 | 21 | 22 | 20 | 17 | 21 | 19 | 108 | 103 | 349
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Laos | 31 | 33 | 33 | 32 | 32 | 30 | 32 | 197 | 197 | 617
Strongyloides stercoralis infection intensity [Count of Participants; unit: Participants] — Population: In phase 2a, the analysis population is the intention-to-treat population, excluding participants lost to follow-up. In phase 2b, the analysis population includes all randomized participants.
  Participants
    number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 197 | 197 | 603
    Light | 6 | 4 | 6 | 3 | 5 | 3 | 4 | 47 | 53 | 131
    Moderate | 13 | 13 | 14 | 12 | 12 | 13 | 12 | 85 | 83 | 257
    Heavy | 11 | 12 | 12 | 14 | 13 | 14 | 13 | 65 | 61 | 215

OUTCOME MEASURES:

1. Primary Outcome: Observed Cure Rate Against Strongyloides Stercoralis
Description: The conversion from being larvae positive pre-treatment to larvae negative post-treatment, or cure rate (CR).
Time Frame: Phase 2a: 21-28 days after treatment; phase 2b: 14-21 days after treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
percentage of participants | 73.3 [54.1 to 87.7] | 89.7 [72.6 to 97.8] | 84.4 [67.2 to 94.7] | 82.8 [64.2 to 94.2] | 96.6 [82.2 to 99.9] | 87.1 [70.2 to 96.4] | 13.8 [3.9 to 31.7] | 92.7 [88.1 to 96.0] | 92.6 [87.9 to 95.9]

2. Secondary Outcome: Observed Larvae-reduction Rate (LRR) Against Strongyloides Stercoralis
Description: Larvae per gram (LPG) stool sample will be assessed by calculating the mean of the larvae counts from the three duplicate Baermann assays and divided by the mean weighted amount of these stool samples. The LRR will be calculated following: (LRR = (1-(mean at follow-up/mean at baseline))*100)
Time Frame: Phase 2a: 21-28 days after treatment; phase 2b: 14-21 days after treatment
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Groups:
- Phase 2a - Arm A (Moxidectin 6 mg): 6 mg Moxidectin at day 0 administered orally
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm A (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
percent change | 98.4 [93.7 to 99.9] | 99.4 [98.1 to 100] | 99.8 [99.3 to 100] | 97.8 [93.2 to 99.9] | 98.6 [95.1 to 100] | 98.5 [95.6 to 99.9] | 27.0 [-2.2 to 48.3] | 99.6 [99.1 to 100] | 99.9 [99.8 to 100]

3. Secondary Outcome: Observed CRs Against Concomitant Soil-transmitted Helminth Infections - Ascaris Lumbricoides
Description: CRs will be calculated for Ascaris lumbricoides infections as described in primary outcome.
Time Frame: Phase 2a: 21-28 days after treatment; phase 2b: 14-21 days after treatment
Population: Participants co-infected with A. lumbricoides
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 9 | 6
percentage of participants |  | 0 [0 to 0] | 100 [100 to 100] | 100 [100 to 100] | 100 [100 to 100] | 0 [0 to 0] |  | 100 [100 to 100] | 83.3 [40.5 to 100]

4. Secondary Outcome: Observed CRs Against Concomitant Soil-transmitted Helminth Infections - Trichuris Trichiura
Description: CRs will be calculated for Trichuris trichiura infections as described in primary outcome.
Time Frame: Phase 2a: 21-28 days after treatment; phase 2b: 14-21 days after treatment
Population: Number of Participants co-infected with T. trichiura
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 1 | 1 | 2 | 10 | 17
percentage of participants | 100 | 100 | 50 | 33 | 0 | 0 | 0 | 100 | 100

5. Secondary Outcome: Observed CRs Against Concomitant Soil-transmitted Helminth Infections - Hookworm
Description: CRs will be calculated for Hookworm infections as described in primary outcome.
Time Frame: Phase 2a: 21-28 days after treatment; phase 2b: 14-21 days after treatment
Population: Participants co-infected with Hookworm
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 17 | 18 | 21 | 17 | 20 | 21 | 17 | 94 | 97
percentage of participants | 0 | 11 | 14 | 0 | 10 | 29 | 0 | 31.9 | 17.5

6. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: Subjects will be kept for observation for at least 3 hours following treatment for any acute AEs. If there is any abnormal finding, the local study physician will perform a full clinical, physical and biochemical examination and findings will be recorded. An emergency kit will be available on site to treat any medical conditions that warrant urgent medical intervention. In addition patients will also be interviewed 2-3 and 24 hours and again 3-4 (phase 2a) or 2-3 (phase 2b) weeks after treatment about the occurrence of AEs. A standardized symptom questionnaire is used, that includes the recording of headache, abdominal pain, itching, nausea, vomiting, diarrhea, allergic reaction as well as any further mentioned event by the participant.
Time Frame: 2-3 hours, 24 hours, and retrospectively 21-28 days (phase 2a) or 14-21 days (phase 2b Arm A and Arm B) after treatment.
Population: Phase 2a: Analysis population N=209 at all time points. Phase 2b: Analysis population at 2-3 hours after drug administration: N=394. Analysis population at 24 hours after drug administration: N=394. Analysis population at 14-21 days after drug administration: N=381.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 197 | 197
Participants
  2-3 hours: Headache | 1 | 1 | 1 | 1 | 2 | 0 | 5 | 11 | 9
  2-3 hours: Abdominal pain | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 12 | 10
  2-3 hours: Itching | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 4
  2-3 hours: Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
  2-3 hours: Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  2-3 hours: Diarrhea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  2-3 hours: Allergic reaction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  24 hours: Headache | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 12
  24 hours: Abdominal pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 21
  24 hours: Itching | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3
  24 hours: Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  24 hours: Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 6
  24 hours: Diarrhea | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  24 hours: Allergic reaction | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  21-28/14-21 days: Headache: number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
  21-28/14-21 days: Headache | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 8 | 1
  21-28/14-21 days: Abdominal pain: number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
  21-28/14-21 days: Abdominal pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 5
  21-28/14-21 days: Itching: number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
  21-28/14-21 days: Itching | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 9 | 1
  21-28/14-21 days: Nausea: number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
  21-28/14-21 days: Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  21-28/14-21 days: Vomiting: number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
  21-28/14-21 days: Vomiting | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  21-28/14-21 days: Diarrhea: number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
  21-28/14-21 days: Diarrhea | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 2
  21-28/14-21 days: Allergic reaction: number analyzed (Participants) | 30 | 29 | 32 | 29 | 30 | 30 | 29 | 192 | 189
  21-28/14-21 days: Allergic reaction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

7. Secondary Outcome: Maximum Concentration (Cmax) of Moxidectin in Adults
Description: Upon oral intake moxidectin levels in blood will be quantified with time using a micro sampling device. Moxidectin will be quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Drug concentrations will be calculated by interpolation from a calibration curve with a foreseen limit of quantification of approximately 5 ng/ml. The PK analysis will be undertaken fitting a structural compartmental PK model.
Time Frame: 0, 2, 4, 6, 7, 24, and 72 hours, and 28 days after treatment.
Population: Data were only collected in phase 2a - Arm D (Moxidectin 8 mg).
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0
ng/mL |  |  |  | 86.1 [76.7 to 89.5] |  |  |  |  |

8. Secondary Outcome: Time to Reach Cmax (Tmax) of Moxidectin in Adults
Description: as for outcome 7
Time Frame: 0, 2, 4, 6, 7, 24, and 72 hours, and 28 days after treatment.
Population: Data were only collected in phase 2a - Arm D (Moxidectin 8 mg).
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0
hours |  |  |  | 4 [4 to 4] |  |  |  |  |

9. Secondary Outcome: Area Under the Curve (AUC) of Moxidectin in Adults
Description: as for outcome 7
Time Frame: 0, 2, 4, 6, 7, 24, and 72 hours, and 28 days after treatment.
Population: Data were only collected in phase 2a - Arm D (Moxidectin 8 mg).
Measure: Median (Inter-Quartile Range); unit: ng/mL*h
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0
ng/mL*h |  |  |  | 5028 [4286 to 5578] |  |  |  |  |

10. Secondary Outcome: Elimination Half Life (T1/2) of Moxidectin in Adults
Description: as for outcome 7
Time Frame: 0, 2, 4, 6, 7, 24, and 72 hours, and 28 days after treatment.
Population: Data were only collected in phase 2a - Arm D (Moxidectin 8 mg).
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
Number analyzed (Participants) | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0
hours |  |  |  | 666 [562 to 759] |  |  |  |  |

ADVERSE EVENTS:
Time Frame: 21-28 days (phase 2a) / 14-21 days (phase 2b)
Description: Participants were monitored at the site for 3 hours following treatment. In addition, participants were interviewed at 2-3 and 24 hours after treatment and retrospectively at 21-28 days (phase 2a) or 14-21 days (phase 2b) about the occurrence of adverse events.
Arm/Group | Phase 2a - Arm A (Moxidectin 2 mg) | Phase 2a - Arm B (Moxidectin 4 mg) | Phase 2a - Arm C (Moxidectin 6 mg) | Phase 2a - Arm D (Moxidectin 8 mg) | Phase 2a - Arm E (Moxidectin 10 mg) | Phase 2a - Arm F (Moxidectin 12 mg) | Phase 2a - Arm G (Placebo) | Phase 2b - Arm A (Moxidectin) | Phase 2b - Arm B (Ivermectin)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33 | 0/33 | 0/32 | 0/32 | 0/30 | 0/32 | 0/197 | 0/197
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33 | 0/33 | 0/32 | 0/32 | 0/30 | 0/32 | 0/197 | 0/197
Other Adverse Events (participants affected / at risk) | 3/31 | 6/33 | 3/33 | 5/32 | 7/32 | 1/30 | 12/32 | 59/197 | 60/197
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2a - Arm A (Moxidectin 2 mg) (N=31) | Phase 2a - Arm B (Moxidectin 4 mg) (N=33) | Phase 2a - Arm C (Moxidectin 6 mg) (N=33) | Phase 2a - Arm D (Moxidectin 8 mg) (N=32) | Phase 2a - Arm E (Moxidectin 10 mg) (N=32) | Phase 2a - Arm F (Moxidectin 12 mg) (N=30) | Phase 2a - Arm G (Placebo) (N=32) | Phase 2b - Arm A (Moxidectin) (N=197) | Phase 2b - Arm B (Ivermectin) (N=197)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 41 (45) | 34 (36)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 6 (6)
Headache (General disorders) | 3 (3) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 1 (1) | 8 (8) | 25 (26) | 21 (22)
Nausea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (8) | 2 (2)
Allergic reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 15 (16) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT04056325/Prot_SAP_000.pdf